CLINICAL TRIAL: NCT02285244
Title: A Phase 2 Feasibility Study of Sotrastaurin for Relapsed and Refractory CLL/SLL/PLL/RT
Brief Title: Sotrastaurin Acetate in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia, Small Lymphocytic Leukemia, Prolymphocytic Leukemia, or Richter's Transformation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision made by the Principal Investigator
Sponsor: James Blachly (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, James Blachly, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-14026; NCI-2014-02002 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COEB071XUS01T
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Prolymphocytic Leukemia; Recurrent Mantle Cell Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Richter Syndrome
MeSH Terms: conditions — Leukemia, Prolymphocytic; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — sotrastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (sotrastaurin acetate) (Experimental): Patients receive sotrastaurin acetate PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sotrastaurin acetate; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sotrastaurin acetate — Given PO
  Other Names: AEB 071; AEB071
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well sotrastaurin acetate works in treating patients with chronic lymphocytic leukemia, small lymphocytic leukemia, prolymphocytic leukemia, or Richter's transformation that has returned or that does not respond to treatment. Sotrastaurin acetate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective clinical response rate of AEB071 (sotrastaurin acetate) treatment in patients with relapsed or refractory chronic lymphocytic leukemia (CLL)/small lymphocytic leukemia (SLL)/prolymphocytic leukemia (PLL)/Richter's transformation (RT).

SECONDARY OBJECTIVES:

I. To determine the feasibility and tolerability of long-term administration of a fixed dose of AEB071 in patients with relapsed or refractory CLL/SLL/PLL.

II. To examine select downstream pharmacodynamic effects in this population of patients after receiving AEB071 including assessment of the wingless-type MMTV integration site family (WNT) signaling pathway.

III. To determine the feasibility and tolerability of AEB071 treatment in patients with relapsed or refractory mantle cell lymphoma (MCL) as well as to gain preliminary data regarding efficacy in this patient population.

TERTIARY OBJECTIVES:

I. Determine the proportion of patients with select germline and somatic deoxyribonucleic acid (DNA) alterations, including in the B-cell receptor (BCR) pathway.

II. Determine how mutational and transcriptional status in key genes affects response to this therapy and may have affected response to prior therapies.

OUTLINE:

Patients receive sotrastaurin acetate orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then at least every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Life expectancy >= 2 months
* Appropriate histologic diagnosis (a) or (b):

  * (a) Histologically documented diagnosis of intermediate or high risk CLL/SLL, B-PLL, and RT arising from CLL/SLL according to the 2008 guidelines, meeting criteria for active disease requiring treatment:

    * Evidence of marrow failure as manifested by the development or worsening of anemia or thrombocytopenia (not attributable to autoimmune hemolytic anemia or thrombocytopenia)
    * Massive (>= 6 cm below the costal margin), progressive or symptomatic splenomegaly
    * Massive nodes (>= 10 cm) or progressive or symptomatic lymphadenopathy
    * Autoimmune anemia and/or thrombocytopenia that is poorly responsive to standard therapy
    * Constitutional symptoms including any of the following:

      * Unintentional weight loss of 10% or more within 6 mos.
      * Significant fatigue limiting activity
      * Fevers >= 100.5 degrees F for 2 weeks or more without evidence of infection
      * Night sweats > 1 month without evidence of infection
    * Need for cytoreduction prior to stem cell transplantation
  * (b) Pathologically documented MCL [defined as either t(11;14) or overexpression of cyclin D1] for the MCL pilot study
* Relapsed after or refractory to at least one prior therapy
* Willingness to undergo all study-related evaluations and procedures
* Ability to understand and willingness to execute a written informed consent document

Exclusion Criteria:

* Prior therapy as follows:

  * Major surgery within 2 weeks
  * Corticosteroids greater than 20 mg/day prednisone (or equivalent) within 2 weeks unless used by inhalation or topical route, or unless necessary for premedication before iodinated contrast dye, or for autoimmune hemolytic anemia
  * Cytotoxic chemotherapy or biologic therapy within 4 weeks, excepting BCR kinase inhibitors for which no wash out is required, or
  * Nitrosoureas within the 6 weeks of the planned first dose of the study drug
* Failure to recover toxicity from prior chemo- or radiotherapy to grade 1
* Known active leukemia or lymphoma of the central nervous system (CNS) requiring therapy
* Inadequate bone marrow function/hematopoietic reserve, except in the case of documented bone-marrow involvement: absolute neutrophil count (ANC) < 1 x 10^9/L
* Inadequate bone marrow function/hematopoietic reserve, except in the case of documented bone-marrow involvement: platelets < 30 x 10^9/L
* Serum total bilirubin > 2 x ULN (upper limit of normal)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x ULN, or > 5 x ULN if CLL/lymphoma is present in the liver
* Estimated glomerular filtration rate (GFR) < 30 mL/min
* Patients who are receiving treatment with medications that are known to be strong inducers or inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4/5 (CYP3A4/5) and CYP3A4/5 substrates with QT prolongation risk that cannot be discontinued prior to study entry
* Clinically significant cardiac diseases, including any of the following:

  * History or presence of ventricular tachyarrhythmia
  * Presence of unstable/uncontrolled atrial fibrillation (with ventricular rate > 100 beats per minute [bpm]); patients with stable atrial fibrillation are eligible provided that they do not meet any of the other exclusion criteria
  * Angina pectoris or acute myocardial infarction within 3 months of starting study drug
  * New York Heart Association (NYHA) functional class III or IV heart failure
  * Labile or uncontrolled hypertension
* History of another malignancy that limits survival to less than 2 years in the estimate of the investigator; basal and squamous cell cancers of the skin, or squamous cell carcinoma of the cervix in situ, which were completely resected or otherwise cured, or localized prostate cancer (Gleason < 5) are eligible
* Gastrointestinal dysfunction, including motility or malabsorption syndromes or inflammatory bowel disease which could limit absorption of AEB071
* Known human immunodeficiency virus (HIV) positivity, or active hepatitis B or C infection with detectible viral nucleic acid in the blood; testing for these viruses is not a required part of screening
* Severe systemic infections requiring intravenous antibiotics within the two weeks prior to initiation of AEB071
* Lactating or pregnant
* Women of child-bearing potential or male partners of women of child-bearing potential who will not agree to use highly effective method of contraception throughout the entire study period and for a minimum of 5 terminal half-lives of AEB071 (approximately 36 hours) after the last dose of study drug; highly effective contraception methods include:

  * Total abstinence or
  * Male or female sterilization or
  * Combination of any two of the following (a+b or a+c or b+c):

    * a. Use of oral, injected or implanted hormonal methods of contraception
    * b. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * c. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential
* Any other life-threatening illness or medical condition that, in the opinion of the investigator, could compromise the safety of the patient or interfere with analysis of study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03-12 (Actual); Primary Completion 2015-03-12 (Actual); Study Completion 2015-03-12 (Actual)

PRIMARY OUTCOMES:
Proportion of CLL/SLL/PLL/RT patients who achieve an objective clinical response, estimated by the number of complete, partial, or partial responses with lymphocytosis divided by the total number of evaluable patients | Up to 9 months
  Categories of response for CLL and PLL patients defined according to criteria published by the International Workshop on CLL. Response for SLL/RT patients will be according to revised response criteria for malignant lymphoma. The objective response rate for all evaluable patients in the phase II study will be calculated with an exact 95% binomial confidence interval (assuming that the number of patients who respond is binomially distributed).

SECONDARY OUTCOMES:
Response duration | From the time at which criteria for CR, PR, or PR with lymphocytosis is first assessed until the date at which recurrent or progressive disease or death due to disease is documented, assessed up to 3 years
  For CLL and PLL patients, defined according to the criteria published by the International Workshop on CLL with the modification outlined by Cheson et al. For SLL/RT patients, responses will be according to revised response criteria for malignant lymphoma. Summarized using standard Kaplan-Meier methods.
Progression free survival (PFS) | Time from the first dose of the study drug until disease progression or death from any cause, assessed up to 3 years
  For CLL and PLL patients, defined according to the criteria published by the International Workshop on CLL with the modification outlined by Cheson et al. For SLL/RT patients, responses will be according to revised response criteria for malignant lymphoma. Summarized using standard Kaplan-Meier methods.
Overall survival (OS) | Time from the first dose of the study drug until death, assessed up to 3 years
  For CLL and PLL patients, defined according to the criteria published by the International Workshop on CLL with the modification outlined by Cheson et al. For SLL/RT patients, responses will be according to revised response criteria for malignant lymphoma. Summarized using standard Kaplan-Meier methods.
Rate of objective clinical response (CR, PR) (optional PLCG2 enriched cohort, if activated) | Up to 3 years
  For CLL and PLL patients, defined according to the criteria published by the International Workshop on CLL with the modification outlined by Cheson et al. For SLL/RT patients, responses will be according to revised response criteria for malignant lymphoma. Summarized using standard Kaplan-Meier methods.
Response duration (optional PLCG2 enriched cohort, if activated) | From the time at which criteria for CR, PR, or PR with lymphocytosis is first assessed until the date at which recurrent or progressive disease or death due to disease is documented, assessed up to 3 years
  For CLL and PLL patients, defined according to the criteria published by the International Workshop on CLL with the modification outlined by Cheson et al. For SLL/RT patients, responses will be according to revised response criteria for malignant lymphoma. Summarized using standard Kaplan-Meier methods.
PFS (optional PLCG2 enriched cohort, if activated) | Time from the first dose of the study drug until disease progression or death from any cause, assessed up to 3 years
  For CLL and PLL patients, defined according to the criteria published by the International Workshop on CLL with the modification outlined by Cheson et al. For SLL/RT patients, responses will be according to revised response criteria for malignant lymphoma. Summarized using standard Kaplan-Meier methods.
OS (optional PLCG2 enriched cohort, if activated) | Time from the first dose of the study drug until death, assessed up to 3 years
  For CLL and PLL patients, defined according to the criteria published by the International Workshop on CLL with the modification outlined by Cheson et al. For SLL/RT patients, responses will be according to revised response criteria for malignant lymphoma. Summarized using standard Kaplan-Meier methods.
Rate of objective clinical response (CR, PR) (MCL cohort) | Up to 3 years
  Responses are defined according the revised response criteria for malignant lymphoma. Summarized using standard Kaplan-Meier methods.
Response duration (MCL cohort) | From the time at which criteria for CR, PR, or PR with lymphocytosis is first assessed until the date at which recurrent or progressive disease or death due to disease is documented, assessed up to 3 years
  Responses are defined according the revised response criteria for malignant lymphoma. Summarized using standard Kaplan-Meier methods.
PFS (MCL cohort) | Time from the first dose of the study drug until disease progression or death from any cause, assessed up to 3 years
  Responses are defined according the revised response criteria for malignant lymphoma. Summarized using standard Kaplan-Meier methods.
OS (MCL cohort) | Time from the first dose of the study drug until death, assessed up to 3 years
  Responses are defined according the revised response criteria for malignant lymphoma. Summarized using standard Kaplan-Meier methods.
Incidence of adverse events (AEs), assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 criteria | Up to 30 days post-treatment
  For each disease group, frequency and severity of adverse events will be collected and summarized by descriptive statistics.
Frequency of AEs requiring dose reduction or drug discontinuation | Up to 30 days post-treatment
  Number of patients who require dose modifications and/or dose delays will be assessed.
Number of courses completed | Up to 30 days post-treatment
  Number of courses started/completed and the reasons for going off-treatment will be assessed.
Pharmacodynamic modulation of the downstream targets of the BCR (including LCP1) after sotrastaurin acetate treatment | Baseline to up to course 1 day 29
  Markers will be summarized univariately in a quantitative manner and also summarized by clinical outcome group graphically to assess potential patterns and relationships. Changes in BCR signaling over time may be evaluated quantitatively using repeated measures models and graphically with individual time plots or box plots.
Pharmacodynamic modulation of the downstream targets of nuclear transcription factor kappa-B after sotrastaurin acetate treatment | Baseline to up to course 1 day 29
  Markers will be summarized univariately in a quantitative manner and also summarized by clinical outcome group graphically to assess potential patterns and relationships.
Pharmacodynamic modulation of downstream targets of WNT/beta-catenin pathway | Baseline to up to course 1 day 29
  Markers will be summarized univariately in a quantitative manner and also summarized by clinical outcome group graphically to assess potential patterns and relationships.
Genomic features associated with response by deep sequencing panel targeted at recurrent mutations in CLL | Up to course 1 day 29
  Markers will be summarized univariately in a quantitative manner and also summarized by clinical outcome group graphically to assess potential patterns and relationships.

CONTACTS AND LOCATIONS:
Overall Officials: James Blachly, MD, Principal Investigator — Ohio State University

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu